CLINICAL TRIAL: NCT02279433
Title: A Phase 1/1B Multi-Center, Non Randomized, Open-Label, Multiple Dose First-In-Human Study Of DS-6051b, An Oral ROS1 And NTRK Inhibitor, In Subjects With Metastatic and/or Unresectable Solid Tumors
Brief Title: A First-in-human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of DS-6051b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Collaborators: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS6051-A-U101
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors
Keywords: Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Neuroendocrine Tumors; Pancreatic Neoplasms
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Neuroendocrine Tumors; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS-6051b (Experimental): DS-6051b is orally administered as 50 mg and 200 mg capsules once daily on Days 1 to 21 of a 21-day cycle. Dose escalation in Part 1 will continue until tentative Recommended Part 2 Dose (RP2D) is determined. In Part 2 participants will receive the RP2D.
  Interventions: Drug: DS6051b

INTERVENTIONS:
Drug: DS6051b — DS-6051b 50 mg and 200 mg capsules for oral administration
  Other Names: Investigational product; DS-6051a (a free base of 6051b)

SUMMARY:
DS-6051b is an orally administered inhibitor of the tyrosine kinases (ROS1) and neurotropic tyrosine kinase receptors (NTRK). This phase 1 first-in-human study evaluates safety and tolerability of DS-6051b in cancer subjects and identify a recommended phase 2 dose (RP2D). In addition, this study will also assess the pharmacokinetic (PK)/pharmacodynamic (PD) profiles and preliminary efficacy of DS-6051b.

DETAILED DESCRIPTION:
The Dose Escalation part (Part 1) of this study will evaluate safety and tolerability, and determine the tentative RP2D. Plasma exposure of DS-6051a and the exposure - QT interval prolongation relationship will also be assessed. Approximately 30 subjects with advanced solid tumors harboring ROS1 or NTRK1, NTRK2, or NTRK3 rearrangement, neuroendocrine carcinoma, or with advanced solid tumors and tumor-induced pain will be enrolled.

The Food Effect (FE) part of this study is to determine the effect of food on the PK of DS-6051a following administration of a single oral dose of DS-6051b. The safety and tolerability of DS-6051b administered with or without food will also be assessed.

After the safety profile of DS-6051b is adequately evaluated, the Dose Expansion part (Part 2) will be initiated to further assess the safety and tolerability, and preliminarily evaluate the efficacy of DS-6051b at the tentative RP2D. Approximately 40 cancer subjects carrying a ROS1 or NTRK1, NTRK2, or NTRK3 rearrangement will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced solid tumors that have relapsed from or are refractory to standard treatment or for which no standard treatment is available
2. Part 1 Dose Escalation subjects must meet 1 of the following criteria:

   * Solid tumors with documented ROS1, NTRK1, NTRK2, or NTRK3 rearrangement
   * Neuroendocrine tumors
   * Solid tumors with tumor-induced pain
3. Part 2 Dose Expansion subjects must meet 1 of the following criteria:

   * NSCLC with documented ROS1, NTRK1, NTRK2, or NTRK3 rearrangement
   * k-RAS wild-type CRC with documented NTRK1, NTRK2, or NTRK3 rearrangement
   * Other solid tumors with documented ROS1, NTRK1, NTRK2, or NTRK3 rearrangement
   * Pulmonary LCNEC;
4. Male or female ≥18 years of age
5. Eastern Cooperative Oncology Group performance status 0 to 1
6. Adequate organ function
7. Adequate blood clotting function
8. Women of childbearing potential must have a negative pregnancy test
9. Willingness to provide archival tumor samples
10. Other inclusion criteria may apply

Exclusion Criteria:

1. Hematological malignancies
2. Known positive HIV infection, or active hepatitis B or C infection
3. Comorbidity that would interfere with therapy
4. Receipt of an allogeneic bone marrow or allogeneic stem cell transplant
5. Concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor
6. History of myocardial infarction and unstable angina within 6 months before study drug treatment; symptomatic congestive heart failure (Congestive Heart Failure New York Heart Association Class III or IV); congenital long QT syndrome; or ventricular arrhythmias defined as grade ≥2 according to NCI CTCAE, v4
7. Clinically active primary central nervous system tumors or brain metastases with the exception of subjects with glioblastoma multiform that carry ROS1 rearrangement
8. Unresolved toxicities from previous anticancer therapy
9. Systemic treatment with anticancer therapy within 3 weeks before study drug treatment
10. Therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment
11. Participation in a therapeutic clinical study within 3 weeks for biological treatments, and within 2 weeks or 5 half-lives, whichever is longer, for small molecule agents, before study drug treatment
12. Concomitant treatment with strong inhibitors or inducers of CYP3A4 and P-glycoprotein
13. Clinically significant malabsorption syndrome or other gastrointestinal disease that would impact drug absorption
14. QTcF values higher than 450 ms at screening
15. Breastfeeding
16. Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose-limiting toxicities | within 21 days following the first dose of treatment
Tumor response | up to 2 years
  Tumor response will be assessed using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for DS-6051a | At Days 1 and 15 of Cycle 1 (21 days)
Time to maximum concentration (Tmax) for DS-6051a | At Days 1 and 15 of Cycle 1 (21 days)
Area under the concentration-time curve from time zero to t (AUC0-t) for DS-6051a | At Days 1 and 15 of Cycle 1 (21 days)
Change from baseline in QTc interval | within 2 years
  ECGs performed to assess QTc interval (ms) at baseline and on study treatment and at the end of treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Oncology, Study Director — AnHeart Therapeutics Inc.
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Chao Family Comprehensive Cancer Center of, Orange, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - New York University, New York, New York
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No